CLINICAL TRIAL: NCT00032565
Title: CSP #476SM - Enhancing Quality of Informed Consent (EQUIC-SM) Self-Monitoring
Brief Title: EQUIC-SM: Enhancing Quality of Informed Consent
Acronym: EQUIC
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Lavori, Philip - Study Chair, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: 476SM
Record Dates: First submitted 2002-03-27; First posted 2002-03-28 (Estimated); Last update posted 2010-09-24 (Estimated); Status verified 2010-09

CONDITIONS: Healthy; Informed Consent

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: No intervention. Telephone interview.

SUMMARY:
Patients in 'parent' cooperative studies projects are interviewed about their experiences in the informed consent process.

DETAILED DESCRIPTION:
Intervention: Self-Monitoring Questionnaire (a questionnaire relating to the process of IC self-administered by study coordinators) and evaluation of the informed consent process using the Brief Informed Consent Evaluation Protocol (BICEP) developed during the EQUIC-DP phase.

Primary Hypothesis: We hypothesize that by focusing attention on what may have become a routinized process, the quality of the IC encounter will be enhanced. We will evaluate the success of this intervention by having the patient-subject complete a telephone questionnaire, the BICEP (Brief Informed Consent Evaluation Protocol), after the IC process is completed.

Primary Outcomes: The quality of the informed consent process, as measured by the BICEP (Brief Informed Consent Evaluation Protocol). The BICEP also offers a method to certify informed consent in routine use.

Study Abstract: Enhancing the Quality of Informed Consent Self-Monitoring (EQUIC-SM) is one component of a VA Cooperative Studies Program-wide initiative on informed consent (EQUIC). Its objective is the field testing and iterative improvement of one intervention in the informed consent (IC) process, self monitoring. Self-monitoring involves having the person obtaining IC complete a Self-Monitoring Questionnaire, or SMQ after the IC encounter with a patient-subject being recruited for a participating study. We conceive of the SMQ as an activation device which prompts the person obtaining IC to monitor how he/she conducts the IC encounter. RESEARCH DESIGN: EQUIC-SM will be conducted in conjunction with participating clinical trials of the VA CSP at multiple VAs throughout the country. Patient-subjects will be recruited from among participants in these parent studies. Parent studies will be randomized to SM protocol or to control sites.

METHODOLOGY: Patient-subjects will be informed about EQUIC-SM at the time that they are first presented with information about the parent study. The person obtaining consent will use a scripted description of EQUIC-SM. If the subject agrees, verbal consent for EQUIC-SM will be obtained. The same parent study informed consent process will be used for both the SM protocol and control arms of EQUIC-SM; however in the SM protocol arm, the person obtaining consent will complete the SMQ after the IC process. In both arms, patient-subjects will be asked to complete the BICEP interview after the parent study IC process is completed. FINDINGS: Investigators will use the results of EQUIC-SM to assess the value of the self-monitoring technique in improving the quality of informed consent. The premise is that focusing the attention of the person obtaining informed consent on the IC process will enhance the quality of the IC encounter, and thus of the informed consent obtained.

SIGNIFICANCE: Practitioners of clinical trials have a responsibility to ensure that patients participation in research be informed and voluntary. This responsibility implies that we should strive continuously to improve the effectiveness of methods for informing prospective research volunteers about experimental studies, thereby enhancing the protection of their interests. If the self-monitoring technique tested in EQUIC-SM proves to enhance the quality of informed consent, this technique may be adapted for wider use in conducting clinical trials, thus representing an important step towards this goal.

ELIGIBILITY:
Inclusion Criteria:

Depends on 'parent' study

Exclusion Criteria:

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients in various VA clinics
Sampling Method: Non-Probability Sample
Enrollment: 836 (Actual)
Dates: Start 2002-11; Primary Completion 2007-07 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Interview: Telephone based assessment of informed consent | immediate

CONTACTS AND LOCATIONS:
Overall Officials: Philip Lavori, PhD, Study Chair — VA Palo Alto Health Care System
Locations (22):
- United States (22):
  - VA Medical Center, Birmingham, Birmingham, Alabama
  - Central Arkansas VHS Eugene J. Towbin Healthcare Ctr, Little Rock, No. Little Rock, Arkansas
  - VA Medical Center, Loma Linda, Loma Linda, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - VA Connecticut Health Care System (West Haven), West Haven, Connecticut
  - Atlanta VA Medical and Rehab Center, Decatur, Decatur, Georgia
  - Edward Hines, Jr. VA Hospital, Hines, Illinois
  - VA Medical Center, Lexington, Lexington, Kentucky
  - Southeast Veterans Healthcare System, New Orleans, New Orleans, Louisiana
  - VA Maryland Health Care System, Baltimore, Baltimore, Maryland
  - VA Medical Center, Jamaica Plain Campus, Boston, Massachusetts
  - VA Boston Healthcare System, Brockton Campus, Brockton, Massachusetts
  - John D. Dingell VA Medical Center, Detroit, Detroit, Michigan
  - VA Medical Center, Minneapolis, Minneapolis, Minnesota
  - VA Western New York Healthcare System at Buffalo, Buffalo, New York
  - VA Medical Center, Northport, Northport, New York
  - VA Medical Center, Durham, Durham, North Carolina
  - VA Medical Center, Cincinnati, Cincinnati, Ohio
  - VA Medical Center, Philadelphia, Philadelphia, Pennsylvania
  - VA North Texas Health Care System, Dallas, Dallas, Texas
  - Michael E. DeBakey VA Medical Center (152), Houston, Texas
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia

REFERENCES:
- [Derived] Lavori PW, Wilt TJ, Sugarman J. Quality assurance questionnaire for professionals fails to improve the quality of informed consent. Clin Trials. 2007;4(6):638-49. doi: 10.1177/1740774507085144. PMID 18042573